CLINICAL TRIAL: NCT01372397
Title: Reversal of Obesity Cardiomyopathy After Gastric Bypass
Brief Title: Reversal of Obesity Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0613
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overall purpose of this study is to determine if weight loss is beneficial for obese patients with diastolic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will have obesity and have a BMI > 35kg/m2.
* Subjects must be between the ages of 35 and 65 years, in order to limit the confounding affect of age on our endpoints.

To determine if potential subjects meet these criteria, they will:

1. be interviewed,
2. their clinical charts reviewed, by the research study coordinator and/or the PI, and
3. undergo a history and physical by a physician (Study Day 2). Subjects who are to undergo gastric bypass surgery will be in the intervention arm. They will be matched with control subjects. We will attempt to have no more than one control subject for each gastric surgery subject.

Exclusion Criteria:

* Subjects who have a condition that may masquerade as diastolic heart failure will be excluded (see Research and Design).
* Subjects who are < 35 or > 65 years, > 400lbs (the weight limit of the MRI table) not obese, unstable, not able to lie flat for the imaging studies, not ambulatory, unable to give informed consent, pregnant, lactating, with atrial flutter or fibrillation, current smokers, or who will undergo a different type of bariatric surgery (not Roux-en-Y gastric bypass) will be excluded from participation.
* Those who have evidence of other major systemic diseases (e.g., cancer, significant lung disease, creatinine > 2.0mg/dL, hemoglobin < 10g/dL, and liver function tests twice the normal range) will be excluded.
* Subjects who have > class I hypertension will be excluded. The investigators will exclude patients with an LV ejection fraction < 45% and those with significant pulmonary hypertension (peak artery pressure > 55mmHg).

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are obese with heart failure and will undergo gastric bypass surgery or who have already had gastric bypass surgery.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-05; Primary Completion 2012-04-26 (Actual); Study Completion 2012-04-26 (Actual)

PRIMARY OUTCOMES:
Cardiac function, myocardial fat deposition | the time frame of the study

SECONDARY OUTCOMES:
liver fat metabolism, plasma lipidomics | the time frame of the study

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Peterson, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States